CLINICAL TRIAL: NCT04172649
Title: A Randomized Controlled Study on Acupuncture for Perioperative Pain After Open Radical Prostatectomy
Brief Title: Acupuncture With Press Tack Needles for Perioperative Pain After Open Radical Prostatectomy
Acronym: AcuPro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Martini-Klinik am UKE GmbH (Other)
Collaborators: Seirin Corporation, Shizuoka City, Japan (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AcuPro 09.2019; DRK S00019884 (Registry Identifier: German Clinical Trials Register)
Record Dates: First submitted 2019-11-13; First posted 2019-11-21 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Prostate Cancer; Perioperative Pain
Keywords: prostate cancer; pain management; acupuncture; acupressure
MeSH Terms: conditions — Prostatic Neoplasms; Agnosia | interventions — Acupuncture Therapy; Acupressure

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acu Arm (Experimental): press tack needle acupuncture (ACU) and routine postoperative analgesic care
  Interventions: Other: Acupuncture
- SHAM Arm (Sham Comparator): press tack placebo acupressure (SHAM) and routine postoperative analgesic care
  Interventions: Other: Acupressure
- CONTROL Arm (No Intervention): Patients in the control group will receive only routine postoperative analgesic care

INTERVENTIONS:
Other: Acupuncture — On the day before surgery, patients randomized to the intervention groups will receive routine postoperative analgesic care with application of 6 bilateral press tack needles (diameter of 0.15mm and length of 0.6mm for P-6 and Shenmen, diameter of 0.20mm and length of 1.2mm for SP-6, Seirin New Pyonex, Seirin Corp., Shizuoka City, Japan).
  Arms: Acu Arm
Other: Acupressure — On the day before surgery, patients randomized to the intervention groups will receive routine postoperative analgesic care with application of 6 bilateral press tack placebos (knob without needle, diameter of 0.15mm and length of 0.6mm for P-6 and Shenmen, diameter of 0.20mm and length of 1.2mm for SP-6, Seirin New Pyonex, Seirin Corp., Shizuoka City, Japan).
  Arms: SHAM Arm

SUMMARY:
Acupuncture has been shown in several meta-analyses and clinical studies, in different surgical settings and chronic back pain, to be a safe adjuvant option for postoperative pain treatment. In this study, the investigator hypothesize that acupuncture can decrease postoperative pain intensity and amount of given analgesics, and accelerate recovery of bowel motility, in patients after open radical prostatectomy.

The investigator will also investigate whether or not acupuncture with needle skin penetration is more efficacious than acupressure.

DETAILED DESCRIPTION:
This study will be a randomized, controlled and partially blinded study with three arms: 1) press tack needle acupuncture (ACU) and routine postoperative analgesic care, 2) press tack placebo acupressure (SHAM) and routine postoperative analgesic care, and 3) only routine postoperative analgesic care (CONTROL).

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18-70 years
* Diagnosis with prostate cancer and scheduled for open radical prostatectomy
* Ability and willingness to follow study instructions and complete all required questionnaires during hospitalization and follow-up
* Written informed consent

Exclusion Criteria:

* Inability to understand the terms of this study
* Simultanously participation in other clinical trials possibly influencing primary or secondary endpoints or any acupuncture-related clinical trials within 30 days prior to inclusion

  * Prior surgery within the last three months
  * Received acupuncture within 6 weeks before surgery
  * Known hypersensitivity or fear of acupuncture
  * Known abuse of drugs, medications and alcohol
  * Chronic pain for more than 3 months
  * Continuous opioid analgesic medications for more than 3 days during the 4 weeks prior to surgery

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 126 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pain intensity measured by Numeric Rating Scale (NRS-11) | postoperative day three
  The primary outcome is to check the effects of permanent needle acupuncture at 6 acupuncture points for changing postoperative pain intensity as measured by the Numeric Rating Scale (NRS-11), calculated as area under the curve (AUC).

SECONDARY OUTCOMES:
Cumulative use (sum in mg) of routine postoperative analgesics | postoperative day three
  Cumulative use (sum in mg) of routine postoperative analgesics
Time to first defecation following surgery | postoperative day three
  Time to first defecation following surgery
EQ-5D-5L for quality of life | 7 days after catheter removal
  fill out a questionnaire: According to the website httpp://euroqol.org/eq-5d-instruments/eq-5d-5l-about/ under the tab "User guide 5L", page 5 in a blue box, it states that EQ-5D-5L is not an abbreviation and should be used and quoted as is. The EQ-5D-5L questionnaire measures quality of life based on 5 different levels (no problems, slight problems, moderate problems, severe problems and extreme problems) to each of the following dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression.

CONTACTS AND LOCATIONS:
Overall Officials: Hans Heinzer, Prof., Principal Investigator — Vice Medical Director and Faculty member of Martini-Klinik
Locations (1):
- Martini-Klinik am UKE GmbH, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No